CLINICAL TRIAL: NCT03256188
Title: Interrupting Prolonged Sitting With Activity Feasibility Study
Brief Title: Interrupting Prolonged Sitting With Activity
Acronym: InPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rebecca Hasson, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00117049
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity
Keywords: classroom; prolonged sitting; sedentary time; time-on-task; children
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active classroom (Experimental): Twenty elementary school teachers implemented 10, 3-minute moderate-to-vigorous physical activity breaks (50-75% of heart rate maximum), 5 days per week in their classrooms over a 16-week period.
  Interventions: Behavioral: Active classroom

INTERVENTIONS:
Behavioral: Active classroom — 30 minutes of moderate-to-vigorous physical activity
  Other Names: InPACT classroom

SUMMARY:
This study tested the feasibility of interrupting prolonged sitting with 10, 3-minute activity breaks in elementary school classrooms. Three elementary schools in Southeast Michigan (20 teachers, 500 students) participated in this study.

DETAILED DESCRIPTION:
School environments have historically provided many opportunities for children to be physically active through comprehensive programs, including recess, intramural physical activity clubs, interscholastic sports and physical education. However, with recent cuts to public school funding and an increased emphasis on standardized test scores, schools districts across the country have reduced time allocated for structured physical activity in favor of additional academic instruction time. This is troubling as uninterrupted prolonged sitting time is associated with increased disruptive behavior, lower academic achievement and increased obesity risk in children. As such, developing low-cost, innovative physical activity interventions aimed at improving weight outcomes and cognitive function in children are warranted.

Researchers have targeted the school classroom, where students spend the majority of their time, as a potential intervention site. Classroom-based physical activity interventions have been largely successful at increasing physical activity, improving physical fitness and academic achievement among children. Yet, no intervention to date has been able to produce significant improvements in weight status, in part due to the intensity, duration and frequency of activities employed (i.e., low-to-moderate intensity; 10-30 minutes per session; 1-2 sessions per day). Preliminary evidence from our laboratory suggests intermittent activity breaks performed at a moderate-to-vigorous intensity elicits greater total daily physical activity energy expenditure without subsequent increases in food intake compared to lower intensity activities. Other researchers have confirmed greater reductions in weight and fat mass in response to higher rather than lower intensity physical activities. In addition, short bursts of activity rather than continuous movements more closely mimics children's natural activity patterns in free-living environments. Hence, incorporating intermittent activity breaks of moderate-to-vigorous intensity as an intervention component may increase the likelihood of classroom-based physical activity interventions improving weight outcomes in children.

Implementing intermittent activity breaks in a classroom will require adjustments to both teaching curricula and classroom design. Current teaching curricula promotes sedentary behaviors by requiring children to spend between 6 and 8 hours in seated academic instruction per day. Moreover, current classroom designs (i.e., size of the classroom and interior areas, type of furniture, flooring and room arrangement) optimize student learning and classroom management with little consideration given to physical activity and movement. Yet, simple adjustments to teaching curricula (i.e. coupling physical activity with teacher's existing lessons) and classroom design (e.g. using smart floor planning to restructure spaces in a classroom) can dramatically increase movement and subsequent learning within that space. In partnership with the School of Education and the Taubman College of Architecture & Urban Planning, two traditionally non-health related fields, the overall objectives of this pilot study are to: 1) develop a classroom curriculum and floor plan that promotes movement, learning and positive behavioral outcomes; and 2) test the feasibility of implementing our classroom-based physical activity intervention (Interrupting Prolonged sitting with ACTivity or INPACT) in three elementary schools (20 classrooms) across the state of Michigan. Third thru fifth grade teachers and students from Columbia Elementary, Estabrook Elementary and Anderson Elementary will be recruited to participate in this pilot study with classroom teachers delivering the physical activity intervention.

ELIGIBILITY:
Inclusion Criteria:

* 3rd thru 6th grade students in participating InPACT classrooms

Exclusion Criteria:

* N/A

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity (student) | 16 weeks
  Direct observation via the System for Observing Play and Leisure Activity in Youth (SOPLAY) was used to assess student physical activity intensity and physical activity minutes completed in the classroom.
Moderate-to-vigorous physical activity (teacher) | 16 weeks
  Direct observation via the System for Observing Play and Leisure Activity in Youth (SOPLAY) was used to assess teacher physical activity intensity and physical activity minutes completed in the classroom.

SECONDARY OUTCOMES:
Transition time | 16 weeks
  Transition time was assessed via direct observation and was calculated as the amount of time from when the teacher completed instructions to his/her class to prepare for an activity break to when students started engaging in the activity break.
Time-on-task | 16 weeks
  Time-on-task was assessed via direct observation and was calculated as the percent of students following the directions of the teacher 30 seconds post activity break.
Physical activity enjoyment | 16 weeks
  Teachers distributed the revised Physical Activity Enjoyment Scale (PACES) to their students to assess enjoyment of participating in the activity breaks.
Physical activity confidence | 16 weeks
  Teachers distributed a single-item question from the Physical Activity Self-Efficacy Scale (PASES) to measure physical activity confidence.
Physical activity heart rate | 16 weeks
  Heart rate during physical activity breaks in the classroom was assessed via heart rate monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Hasson, PhD, Principal Investigator — University of Michigan
Locations (1):
- Childhood Disparities Research Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No